CLINICAL TRIAL: NCT00207415
Title: A Comparison of the ASHC and CDSMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCCDPHP-MM0512-03/03; MM0512-03/03
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Arthritis
Keywords: arthritis; self management
MeSH Terms: conditions — Arthritis

INTERVENTIONS:
Behavioral: ASHC and CDSMP

SUMMARY:
The arthritis-specific Arthritis Self Help Course (ASHC) and the more generic Chronic Disease Self Management Program (CDSMP) teach generalizable skills for managing arthritis and other chronic diseases. In some locations it may be more feasible to combine efforts and offer the generic course rather than the arthritis-specific program. However anecdotal evidence has questioned whether people with arthritis obtain as much benefit from the more generic course as they do the arthritis-specific course. The primary purpose of this research study is to compare health outcomes among people with arthritis who participate in either ASHC or the CDSMP. The University of Illinois Project is emphasizing recruiting a balance of uran and rural participants. The results of this research will be used to guide Arthritis program recommendations on the use of ASHC and CDSMP to improve the quality of life for people with arthritis.

ELIGIBILITY:
Inclusion Criteria:

Adult with self reported arthritis-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Health status at 6 month follow up
Health Care utilization at 6 month follow up

SECONDARY OUTCOMES:
self management behaviors at 6 month follow up
self efficacy at 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mary Brown, MD, MPH, Principal Investigator — University of Illinois College of Medicine Rockford